CLINICAL TRIAL: NCT05949346
Title: Treatment Efficacy of Multiple Family Narrative Therapy for Chinese Families of Children With Dyslexia: a Randomized Controlled Trial
Brief Title: Multiple Family Narrative Therapy for Chinese Families of Children With Dyslexia
Acronym: MFNT-CDYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: University Grants Committee, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RGC Ref No. 12607921; General Research Fund (GRF) (Other Grant/Funding Number: University Grants Committee (UGC))
Record Dates: First submitted 2023-07-09; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2021-03

CONDITIONS: Dyslexia; Special Education; Special Needs Children
Keywords: Dyslexia; Narrative therapy; Efficacy; Intervention; Multiple family group; Parent-child; Special educational needs
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MFNT Intervention (Treatment Group) (Experimental): Parents of children with dyslexia who are randomized in Treatment Group will first take part in a pre-tested 4-session MFNT intervention programme. The parents will participate in lectures, group discussions, video demonstrations, and in-group exercises offered in these four mentored sessions, while their children will attend the second and fourth sessions.
  Interventions: Behavioral: Multiple Family Narrative Therapy (MFNT)
- MFNT Intervention (Wait Listing Control Group) (Experimental): Families of children with dyslexia who are randomized in Wait Listing Control Group receive services as usual by the school personnel during the intervention period. The 4-session MFNT intervention program will be delivered to them after the intervention period.
  Interventions: Behavioral: School services for families of children with Dyslexia

INTERVENTIONS:
Behavioral: Multiple Family Narrative Therapy (MFNT) — MFNT consist of 4 weekly group sessions with selected themes from both multiple family therapy (MFT) and narrative therapy (NT) offered in a group format. The family is treated as a system through both psychodynamic practices and attachment theories to manage symptoms, to achieve family resilience, and to empower both parents and child to share their unique and lived value-driven experiences. MFNT provides families with therapeutic environments that are conducive to learning and modelling in order to facilitate the process of building healthier parent-child dyads.
  Arms: MFNT Intervention (Treatment Group)
Behavioral: School services for families of children with Dyslexia — Selected school personnel will deliver services as usual for the control group.
  Arms: MFNT Intervention (Wait Listing Control Group)

SUMMARY:
The goal of this randomized controlled trial (RCT) is to develop and to implement a multiple family narrative therapy (MFNT) intervention consisting of parent-child relationships training among Chinese families of children with Dyslexia (CFCDs). The intervention aims to reduce the psychological distress of parents and their child, thus improving parent-child relationships, and the trial aims to assess the effectiveness of MFNT among them. A RCT design supplemented by qualitative interviews will be used to evaluate the effectiveness of MFNT on family welfare.

DETAILED DESCRIPTION:
Dyslexia is a learning disability that causes problems with reading, writing, sequential learning, and phonological processing. It is a diagnosable disorder that commonly coexist with attention-deficit and hyperactivity disorder (ADHD). The estimated percentage of dyslexia in Hong Kong ranges from 9.7 to 12.6%. From 2016 to 2019, the number of students with special learning difficulties in both primary and secondary schools increased by 8.3%. These current statistics project that the number of children with dyslexia will continue to rise in the near future.

International studies indicated that dyslexia impacts the whole family. There are three common problems experienced by families of children with dyslexia: 1) problematic parent-child relationship; 2) parental and psychological distress; and 3) lack of social support. Statistics in Hong Kong also show that Chinese families of children with dyslexia experience similar problems. With daily academic demands, parents are constantly looking for effective ways to manage problems faced by their children with dyslexia even though they do not fully understand their child's dyslexia conditions. In Hong Kong, few studies of psychoeducational models have focused on parent-child relationships, parental stress, and social support for families of children with learning disabilities. The psychological approaches mainly address the behavioural changes of children with Special Educational Needs (SEN). To offset this research gap, it is important to adopt a psychoeducational model and evaluate the effects of the model's intervention on both parents and their children with SEN.

This study addresses a need in the Hong Kong Chinese community and has four expected outcomes: 1) it tests the effectiveness of Multiple Family Narrative Therapy (MFNT) as a brief-targeted intervention model; 2) it facilitates a participatory approach that engages both parents and children; 3) it designs a practice manual that is culturally applicable in the Chinese context; and 4) it encourages the use of the practice manual that outlines a tested model in school and integrative family services.

This study is an evidence-informed and knowledge-building study that aims to test the effectiveness of a brief-targeted MFNT integrative family therapy in Hong Kong compared to a "Treatment as Usual" school-focused approach to work with Chinese family of children with Dyslexia (CFCDs). This approach will target the importance of shifting from academic achievement driven approach, which intensify conflictual parent-child relationship to a collaborative model where family members can review one's identity and re-choose the pattern of interaction among the family members.

The first objective of this study is to test the effectiveness of a brief-targeted Multiple Family Narrative Therapy (MFNT) for Chinese families of children with dyslexia (CFCDs) in Hong Kong, in reducing psychological distress of parents and children, building healthy parent-child relationships, and promoting the use of social support. The second objective is to examine the process of change in attitudes and interactions among family members participating in MFNT.

ELIGIBILITY:
Inclusion Criteria:

* Participants 7-13 years old and their parents
* Dyslexia diagnosis (by psychiatrist or educational psychologist or clinical psychologist)
* Diagnosis with comorbidity of other learning disabilities
* Cantonese speaking participants (child and parents)
* At least one of the parents, but not siblings nor grandparents, can commit to all four sessions
* Participants able to comply with all testing and study requirements

Exclusion Criteria:

* Formal current diagnosis of psychosis
* Limitation in daily communication
* Previous service recipients of Narrative Therapy or Multiple Family Group
* Non-Cantonese speaking child or parent
* Parents or children who refuse to give written consent for their participation in the study

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Kessler Psychological Distress Scale (KPDS) | 1 week prior intervention, Intervention week 4, and 3 months post-intervention
  Kessler Psychological Distress Scale is a 10-item scale completed by the child and the child's parent. It assesses the frequency of distress-related feelings in the past month on a 5-point Likert Scale (1=None of the time; 2=A little of the time; 3=Some of the time; 4=Most of the time; 5=All of the time). The scale is reliable and valid for the local context, given it will be delivered in Chinese. Changes in scores of Kessler Psychological Distress Scale will be evaluated before, after the intervention as well as at a follow-up assessment (3 months after the end of the intervention).
Parental Stress Scale (PSS) | 1 week prior intervention, Intervention week 4, and 3 months post-intervention
  Parental Stress Scale (PSS) consists of 17 items on a 6-point scale (1 = strongly disagree; 2 = disagree; 3= somewhat disagree; 4 = somewhat agree; 5 = agree; 6 = strongly agree) measuring parents' perception of parental stress. Seven items require reverse scoring. A total score is calculated, with higher scores indicating higher levels of parental stress. The Chinese version of the scale has been translated and validated. Changes in its total score will be evaluated before, after the intervention as well as at a follow-up assessment (3 months after the end of the intervention).
Parent-Child Relationship Scale | 1 week prior intervention, Intervention week 4, and 3 months post-intervention
  Parent-Child Relationship Scale is a scale that assesses subjects' perceptions of their current relationship with their children. It consists of 17 items based on 5-point scale, ranging from 1 = never to 5 = always. The scale uses mean score, and a higher score indicates a more positive parent-child relationship. Changes in its mean score will be evaluated before, after the intervention as well as at a follow-up assessment (3 months after the end of the intervention).
Parental Bonding Inventory (PBI) | 1 week prior intervention, Intervention week 4, and 3 months post-intervention
  Parental Bonding Inventory (PBI) is a 25-item instrument assessing levels of parental care and overprotection perceived by the child. It consisted of two subscales termed 'care' and 'overprotection/control'. The measure is to be completed for both mothers and fathers separately, with each parent being scored on a 4-point Likert scale (Very unlike = 0, Moderately unlike = 1, Moderately like = 2, Very like = 3). Changes in the scores in "care" and "overprotection/control" subscales in both father and mother will be evaluated before, after the intervention as well as at a follow-up assessment (3 months after the end of the intervention).

SECONDARY OUTCOMES:
Satisfaction With Family Life Scale (SWFL) | 1 week prior intervention, Intervention week 4, and 3 months post-intervention
  Satisfaction With Family Life Scale (SWFL) is a 5-item scale that assesses an individual's global judgment of family satisfaction. Parents and children were required to agree or disagree with global statements about family life on a 7-point Likert-type scale ranging from 1 = strongly disagree to 7 = strongly agree. This instrument has been successfully used in a variety of family samples and offers a brief, widely applicable tool to measure satisfaction with family life. Changes in its total score will be evaluated before, after the intervention as well as at a follow-up assessment (3 months after the end of the intervention).
Guilt and Shame Questionnaire (GSQ) | 1 week prior intervention, Intervention week 4, and 3 months post-intervention
  Guilt and Shame Questionnaire (GSQ) is a 10-item scale to assess one's feelings of guilt and shame associated with disabilities including but not limited to mental illness. It consisted of two subscale - shame and guilt, both are rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). The scale was completed by parents and children. The evaluation of guilt and shame is calculated based on the sum scores of each subscale. Changes in scores of total scale, guilt and shame subscales will be evaluated before, after the intervention as well as at a follow-up assessment (3 months after the end of the intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Tak Mau Chan, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Department of Social Work, Hong Kong Baptist University, Hong Kong, China, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided